CLINICAL TRIAL: NCT02573675
Title: An Assessment on Current Outcomes of Peritoneal Dialysis in Korea
Acronym: PDKOREA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ewha Womans University (Other)
Responsible Party: Sponsor
Other Study IDs: PDKOREA-1
Record Dates: First submitted 2015-10-08; First posted 2015-10-12 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Kidney Failure, Chronic
Keywords: hemodialysis; peritoneal dialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study, the recent trends in outcomes according to the dialysis modality in Korea since 2009, the effect of the use of peritoneal dialysis solutions containing icodextrin or high-glucose on various outcomes, the usefulness of 'PD first strategy', and the economic burden according to the dialysis modality will be investigated retrospectively using the Korean Health Insurance Review and Assessment Service (HIRA) database.

DETAILED DESCRIPTION:
This study is designed as an observational and retrospective cohort study, thus there will be no intervention or specified prescription.

For the comparison of outcomes according to dialysis modality, we will adopt an intention-to-treat analysis, and consider the dialysis modality at day 90 to be the initial dialysis modality. However, the investigators will also regard the dialysis modality at day 30 as the initial dialysis modality in order to evaluate and compare earlier mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients who started dialysis during the study period and remained on the dialysis therapy for at least 90 days

Exclusion Criteria:

* Patients who were younger than 18 years of age
* Patients who survived for less than 90 days from the date of dialysis initiation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All incident dialysis patients who started chronic dialysis therapy between January 1, 2009 and December 31, 2014 in Korea
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2015-11; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Survival rate according to dialysis modality | up to 5 years

REFERENCES:
- [Background] Kim H, Kim KH, Park K, Kang SW, Yoo TH, Ahn SV, Ahn HS, Hann HJ, Lee S, Ryu JH, Kim SJ, Kang DH, Choi KB, Ryu DR. A population-based approach indicates an overall higher patient mortality with peritoneal dialysis compared to hemodialysis in Korea. Kidney Int. 2014 Nov;86(5):991-1000. doi: 10.1038/ki.2014.163. Epub 2014 May 7. PMID 24805104